CLINICAL TRIAL: NCT04395404
Title: Structural Orbital Changes in Anophthalmic Socket Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: s62697
Record Dates: First submitted 2020-05-11; First posted 2020-05-20 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Anophthalmos; Acquired; Anophthalmic Socket Syndrome
MeSH Terms: conditions — Anophthalmos

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Patients with unilateral ASS, with and without the prosthesis in situ, are analysed by 3D- magnetic resonance imaging (MRI) with 64 channel head coil using T1 and T2 weighted, DIXON/ IDEAL, and T2 inversion recovery sequences.

SUMMARY:
Understand better the aetiology and physiopathogenesis of anophthalmic socket syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Unilateral anophthalmic socket syndrome (superior sulcus grading 0 till 4)
* Enucleation/evisceration with primary implant more than 5 years ago
* After informed consent

Exclusion Criteria:

* MRI absolute and relative contraindications such as metallic fragments or metallic containing devices,
* history of orbital trauma, previous anophthalmic socket and eyelid surgery, inflammation, infection, buphthalmos, congenital anophthalmos and radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Displacement of orbital structures | At least 5 years after enucleation or evisceration
  mm in x,y,z axis
Volumetric orbital difference | At least 5 years after enucleation or evisceration
  ml
Surface comparisson of bony orbits | At least 5 years after enucleation or evisceration
  mm

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No